CLINICAL TRIAL: NCT04945304
Title: 9-Step Magnetic Assisted Conversion From Sleeve Gastrectomy to Roux-en-Y Gastric Bypass and Hiatoplasty by Single-Port.
Brief Title: 9-Step Magnetic Bariatric Revisional Surgery
Status: Recruiting | Type: Observational
Sponsor: Unidad Internacional de Cirugia Bariatrica y Metabolica (Other)
Responsible Party: Principal Investigator, Guillermo Borjas, Director of the International Bariatric and Metabolic Surgery Unit, Unidad Internacional de Cirugia Bariatrica y Metabolica
Other Study IDs: BariatriaInternacional
Record Dates: First submitted 2021-05-31; First posted 2021-06-30 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2022-07

CONDITIONS: Bariatric Surgery Candidate; GERD; Revisional Bariatric Surgery
Keywords: revisional surgery; bariatric surgery; gastric bypass; single port; sleeve gastrectomy; magnetic surgery
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Magnetic bariatric surgery: Bariatric procedure performed in a human using magnetic assistance in the steps of the surgery
  Interventions: Procedure: magnetic bariatric surgery; Procedure: Magnetic gastric bypass

INTERVENTIONS:
Procedure: magnetic bariatric surgery — Perform a roux-en-y gastric bypass, sleeve gastrectomy, nissen-sleeve or revisional bariatric procedure with magnetic assistance
Procedure: Magnetic gastric bypass — Using the magnetic assistance to perform a gastric bypass

SUMMARY:
RYGB represents one of the best alternatives for weight loss in obese patients achieving a weight loss of up to 60% and a resolution of comorbidities of 70%. Revision surgery contemplates multiple techniques including the conversion from one surgical technique to another, structural changes to the primary technique, among others. GERD is now a long-term problem for patients who have undergone LGS. RYGB is one of the best techniques to resolve this problem.

DETAILED DESCRIPTION:
Roux-en-y gastric bypass is performed with the patient in the French position by a bariatric surgeon with 8 years of experience. A single port was placed in the umbilicus, an additional trocar (5mm) was placed in the right side of the abdomen. The surgery is started by performing the liver retraction with the grasper plus magnet attached to the border for the correct visualization of the surgical field. Later, the division of the major curvature of the omentum is started, and as it is performed in a superior direction, the magnet is positioned to retract the fundus and finishing exposing the esophageal hiatus where a hiatal hernia is visualized, which is decided to be repaired transoperatively. For the hiatoplasty, after placing a reference around the stomach, the magnet is positioned in that reference to retract the stomach and esophagus and to be able to suture the hernia defect. Then we proceed to perform the RYGB with the simplified technique, starting with the reference attached to the magnet but this time at the opposite end to start the resection of the lesser omentum, a minor step prior to the confection of the pouch. The pouch confection is done with 3 blue cartridges. Continuing with the procedure, the retraction of the transverse colon is performed with the use of the magnet to visualize the treitz angle and start the 60 cm measurement of the biliopancreatic limb. Later, gastrojejunal anastomosis is performed traditionally. Once this step is finished, the 100 cm alimentary limb is measured and then, the magnet-assisted jejunal anastomosis is performed. The Petersen defect and the intermesenteric defect is closed assisted by magnets. A methylene blue leak test is routinely performed, with negative results, this time testing both anastomoses. Finally, the magnet-assisted omega section is made with the retraction of the limb to finish the Roux-en-Y.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years
* Candidate to bariatric surgery
* Obesity
* BMI Greater than 30 kg/m2

Exclusion Criteria:

* Uncontrolled co-morbidities
* patients with pacemakers, defibrillators, or other electromedical implants
* Abnormal coagulation blood tests
* Patients with hepatic diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients candidates to bariatric surgery in the international unit of bariatric and metabolic surgery
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-05-31 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
complications | 30 days
  adverse surgical events
device malfunction | 1-2 hours
  any adverse event with the magnetic grasper
surgical time | 30 days
  report the surgical time using the magnetic assistance

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Borjas, MD. PhD, Principal Investigator — International Unit of Bariatric and Metabolic Surgery
Locations (1):
- Unidad Internacional de Cirugía Bariátrica y Metabólica, Maracaibo, Zulia, Venezuela

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Guillermo B, Nestor S, Maria G, Ali U, Eduardo R, Andres M. 9-step magnetic assisted conversion from sleeve gastrectomy to roux-en-Y gastric bypass and hiatoplasty by single-port: Case report. Int J Surg Case Rep. 2021 Sep;86:106294. doi: 10.1016/j.ijscr.2021.106294. Epub 2021 Aug 11. PMID 34419721